CLINICAL TRIAL: NCT03225586
Title: Prospective Urban Rural Epidemiology Study
Acronym: PURE
Status: Recruiting | Type: Observational
Sponsor: Population Health Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Principal Investigator, Salim Yusuf's office, Executive Director, Population Health Research Institute, Population Health Research Institute
Other Study IDs: PURE
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Cardiovascular Diseases; Risk Factor, Cardiovascular; Health Behavior; Environmental Exposure; Lung Diseases; Cancer; Injuries; Renal Disease; Communicable Disease
Keywords: Non-communicable Diseases, Risk Factors
MeSH Terms: conditions — Cardiovascular Diseases; Health Behavior; Lung Diseases; Neoplasms; Wounds and Injuries; Kidney Diseases; Communicable Diseases; Noncommunicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, Serum, Plasma, Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults: Between 35 to 70 years of age at time of enrollment

SUMMARY:
To examine the impact of health determinants at the individual (e.g. health related behaviors) and societal level (e.g. environmental factors, health related policy, quality of health systems) on health outcomes (e.g. death, non-communicable disease development) across a range of socioeconomic and health resource settings. Additional components of this study will examine genetic factors for non-communicable diseases. This will be examined both through a cross sectional component, and prospectively (cohort component).

DETAILED DESCRIPTION:
1. To examine the relationship between societal influences and prevalence of risk factors and chronic noncommunicable diseases. Societal determinants are measured by an index of measures from each of the 4 domains of interest: built environment, food and nutrition policy, psychosocial/socioeconomic factors, and tobacco.
2. To examine the relationship between societal determinants and incidence of chronic noncommunicable disease events (e.g. cardiovascular disease, cancer) and on changes in rates of selected risk factors (e.g. smoking)
3. To examine the relationship between health related behaviors (e.g. diet, physical activity, smoking, alcohol) and health outcomes (e.g. death, non-communicable diseases)
4. The quality of health systems across a diverse range of health resource settings, and how this impacts health outcomes
5. Genetic factors for non-communicable diseases

ELIGIBILITY:
Inclusion Criteria:

* consenting adults between 35-70 years of age

Exclusion Criteria:

* none

Ages: 35 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — Both Men and Women
Study Population: Adults aged 35 to 70 years from communities in low-, middle-, and high-income regions of the world representing various levels of development and encompassing great sociocultural diversity.
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2002-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
incident cardiovascular disease | mean follow up of 10 years
  cardiovascular death, stroke, myocardial infarction, heart failure

SECONDARY OUTCOMES:
incident cancer | mean follow up of 10 years
  total and cause specific cancers
Incident COPD | mean follow up of 10 years
  development of COPD
Incident Asthma | mean follow up of 10 years
  development of asthma
Pneumonia | mean follow up of 10 years
  hospitalization for pneumonia
Respiratory outcomes | mean follow up of 10 years
  change in pulmonary function test
All Cause Hospitalizations | mean follow up of 10 years
  All cause hospitalizations
Kidney disease | mean follow up of 10 years
  end stage renal disease, dialysis, transplant, changes in renal function
All cause and cause specific mortality | mean follow up of 10 years
  death from all causes, and cause specific deaths
incident diabetes | mean follow up of 10 years
  development of diabetes
obesity | mean follow up of 10 years
  development of obesity, change in BMI
hypertension | mean follow up of 10 years
  development of hypertension and changes in blood pressure
incident injuries | mean follow up of 10 years
  assessing fatal and non-fatal injuries due road traffic accidents and falls

CONTACTS AND LOCATIONS:
Overall Officials: Salim Yusuf, DPhil, Principal Investigator — Executive Director
Locations (34):
- Estudios Clinicos Latinoamerica ECLA, Rosario, Santa Fe Province, Argentina
- Independent University, Bangladesh, Dhaka, Bangladesh
- Dante Pazzanese Institute of Cardiology, São Paulo, Brazil
- Canada (4):
  - Simon Fraser University, Vancouver, British Columbia
  - Population Health Research Institute, Hamilton, Ontario
  - University of Ottawa, Ottawa, Ontario
  - Université Laval Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec
- Universidad de La Frontera, Temuco, Chile
- State Key Laboratory of Cardiovascular Disease, Fuwai Hospital, Beijing, China
- Fundacion Oftalmologica de Santander - FOSCAL, Floridablanca, Santander Department, Colombia
- India (5):
  - St John's Research Institute, Bangalore, Karnataka
  - Health Action by People, Thiruvananthapuram, Kerala
  - Eternal Heart Care Centre and Research Institute, Jaipur, Rajasthan
  - Madras Diabetes Research Foundation, Chennai, Tamil Nadu
  - Post Graduate Institute of Medical Education and Research (PGIMER), Chandigarh
- Isfahan University of Medical Sciences, Isfahan, Iran
- Research Institute of Cardiology & Internal Diseases, Almaty, Kazakhstan
- Kyrgyz Society of Cardiology, National Center of Cardiology and Internal Disease, Bishkek, Kyrgyzstan
- Malaysia (2):
  - Universiti Teknologi MARA, UCSI Universiti, Kuala Lumpur
  - University Kebangsaan Malaysia, Kuala Lumpur
- Aga Khan University, Karachi, Pakistan
- Birzeit University, Birzeit, Ramallah, Palestinian Territories
- Universidad Peruana Cayetano Heredia, Lima, Peru
- University of Philippines, Section of Adult Medicine & Medical Research Unit, Manila, Philippines
- Wroclaw Medical University & Department of Internal Medicine, Wroclaw, Poland
- Research Institute for Complex Issues of Cardiovascular Diseases, Kemerovo, Russia
- King Saud University, Riyadh, Saudi Arabia
- South Africa (2):
  - School of Public Health, University of the Western Cape, Bellville
  - North-West University, Potchefstroom
- Sahlgrenska University Hospital/Östra Hospital, Gothenburg, Sweden
- Pamoja Tunaweza Women Center, Moshi, Tanzania
- Istanbul Medeniyet University, Istanbul, Turkey (Türkiye)
- Dubai Medical University, Dubai, United Arab Emirates
- University of Zimbabwe College of Health Sciences, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
During study conduct only with the investigators who have participated /contributed to the study. Select summary data may be shared with policy makers for specific purposes.The study exec will consider specific requests for data analyses by non-contributing individuals 3 years after the study has been completed (i.e. complete recruitment and a minimum of 10 years follow up in all) and the participating investigators have had an opportunity to explore questions that they are interested in. Costs related to data curating ,and related efforts will need to be met by anybody not contributing to the study and requesting analyses
Supporting Information: Study Protocol, CSR
Time Frame: complete recruitment and a minimum of 10 years follow up in all
Access Criteria: The study exec will consider specific requests for data analyses by non-contributing individuals 3 years after the study has been completed (i.e. complete recruitment and a minimum of 10 years follow up in all) and the participating investigators have had an opportunity to explore questions that they are interested in.

REFERENCES:
- [Background] Dehghan M, Al Hamad N, Yusufali A, Nusrath F, Yusuf S, Merchant AT. Development of a semi-quantitative food frequency questionnaire for use in United Arab Emirates and Kuwait based on local foods. Nutr J. 2005 May 27;4:18. doi: 10.1186/1475-2891-4-18. PMID 15921524
- [Background] Merchant AT, Dehghan M, Chifamba J, Terera G, Yusuf S. Nutrient estimation from an FFQ developed for a Black Zimbabwean population. Nutr J. 2005 Dec 13;4:37. doi: 10.1186/1475-2891-4-37. PMID 16351722
- [Background] Merchant AT, Dehghan M. Food composition database development for between country comparisons. Nutr J. 2006 Jan 19;5:2. doi: 10.1186/1475-2891-5-2. PMID 16423289
- [Background] Vaz M, Bharathi AV, Thomas T, Yusuf S, Kurpad AV. The repeatability of self reported physical activity patterns in rural South India. Asia Pac J Clin Nutr. 2009;18(1):71-5. PMID 19329398
- [Background] Dehghan M, del Cerro S, Zhang X, Cuneo JM, Linetzky B, Diaz R, Merchant AT. Validation of a semi-quantitative Food Frequency Questionnaire for Argentinean adults. PLoS One. 2012;7(5):e37958. doi: 10.1371/journal.pone.0037958. Epub 2012 May 25. PMID 22662256
- [Background] Dehghan M, Martinez S, Zhang X, Seron P, Lanas F, Islam S, Merchant AT. Relative validity of an FFQ to estimate daily food and nutrient intakes for Chilean adults. Public Health Nutr. 2013 Oct;16(10):1782-8. doi: 10.1017/S1368980012004107. Epub 2012 Sep 21. PMID 22995762
- [Background] Dehghan M, Lopez Jaramillo P, Duenas R, Anaya LL, Garcia RG, Zhang X, Islam S, Merchant AT. Development and validation of a quantitative food frequency questionnaire among rural- and urban-dwelling adults in Colombia. J Nutr Educ Behav. 2012 Nov-Dec;44(6):609-13. doi: 10.1016/j.jneb.2010.10.001. Epub 2011 Jul 7. PMID 21737352
- [Background] Khatib R, Schwalm JD, Yusuf S, Haynes RB, McKee M, Khan M, Nieuwlaat R. Patient and healthcare provider barriers to hypertension awareness, treatment and follow up: a systematic review and meta-analysis of qualitative and quantitative studies. PLoS One. 2014 Jan 15;9(1):e84238. doi: 10.1371/journal.pone.0084238. eCollection 2014. PMID 24454721
- [Result] Teo K, Chow CK, Vaz M, Rangarajan S, Yusuf S; PURE Investigators-Writing Group. The Prospective Urban Rural Epidemiology (PURE) study: examining the impact of societal influences on chronic noncommunicable diseases in low-, middle-, and high-income countries. Am Heart J. 2009 Jul;158(1):1-7.e1. doi: 10.1016/j.ahj.2009.04.019. PMID 19540385
- [Result] Chow CK, Lock K, Teo K, Subramanian SV, McKee M, Yusuf S. Environmental and societal influences acting on cardiovascular risk factors and disease at a population level: a review. Int J Epidemiol. 2009 Dec;38(6):1580-94. doi: 10.1093/ije/dyn258. Epub 2009 Mar 4. PMID 19261658
- [Result] Bharathi AV, Kurpad AV, Thomas T, Yusuf S, Saraswathi G, Vaz M. Development of food frequency questionnaires and a nutrient database for the Prospective Urban and Rural Epidemiological (PURE) pilot study in South India: methodological issues. Asia Pac J Clin Nutr. 2008;17(1):178-85. PMID 18364343
- [Result] Iqbal R, Ajayan K, Bharathi AV, Zhang X, Islam S, Soman CR, Merchant AT. Refinement and validation of an FFQ developed to estimate macro- and micronutrient intakes in a south Indian population. Public Health Nutr. 2009 Jan;12(1):12-8. doi: 10.1017/S1368980008001845. Epub 2008 Mar 7. PMID 18325134
- [Result] Chow CK, Lock K, Madhavan M, Corsi DJ, Gilmore AB, Subramanian SV, Li W, Swaminathan S, Lopez-Jaramillo P, Avezum A, Lear SA, Dagenais G, Teo K, McKee M, Yusuf S. Environmental Profile of a Community's Health (EPOCH): an instrument to measure environmental determinants of cardiovascular health in five countries. PLoS One. 2010 Dec 10;5(12):e14294. doi: 10.1371/journal.pone.0014294. PMID 21170320
- [Result] Mir H, Buchanan D, Gilmore A, McKee M, Yusuf S, Chow CK. Cigarette pack labelling in 12 countries at different levels of economic development. J Public Health Policy. 2011 May;32(2):146-64. doi: 10.1057/jphp.2011.3. Epub 2011 Mar 3. PMID 21368847
- [Result] Yusuf S, Islam S, Chow CK, Rangarajan S, Dagenais G, Diaz R, Gupta R, Kelishadi R, Iqbal R, Avezum A, Kruger A, Kutty R, Lanas F, Lisheng L, Wei L, Lopez-Jaramillo P, Oguz A, Rahman O, Swidan H, Yusoff K, Zatonski W, Rosengren A, Teo KK; Prospective Urban Rural Epidemiology (PURE) Study Investigators. Use of secondary prevention drugs for cardiovascular disease in the community in high-income, middle-income, and low-income countries (the PURE Study): a prospective epidemiological survey. Lancet. 2011 Oct 1;378(9798):1231-43. doi: 10.1016/S0140-6736(11)61215-4. Epub 2011 Aug 26. PMID 21872920
- [Result] Gasevic D, Vukmirovich I, Yusuf S, Teo K, Chow C, Dagenais G, Lear SA. A direct assessment of "obesogenic" built environments: challenges and recommendations. J Environ Public Health. 2011;2011:161574. doi: 10.1155/2011/161574. Epub 2011 Nov 15. PMID 22174727
- [Result] Corsi DJ, Subramanian SV, McKee M, Li W, Swaminathan S, Lopez-Jaramillo P, Avezum A, Lear SA, Dagenais G, Rangarajan S, Teo K, Yusuf S, Chow CK. Environmental Profile of a Community's Health (EPOCH): an ecometric assessment of measures of the community environment based on individual perception. PLoS One. 2012;7(9):e44410. doi: 10.1371/journal.pone.0044410. Epub 2012 Sep 4. PMID 22973446
- [Result] Dehghan M, Ilow R, Zatonska K, Szuba A, Zhang X, Mente A, Regulska-Ilow B. Development, reproducibility and validity of the food frequency questionnaire in the Poland arm of the Prospective Urban and Rural Epidemiological (PURE) study. J Hum Nutr Diet. 2012 Jun;25(3):225-32. doi: 10.1111/j.1365-277X.2012.01240.x. Epub 2012 Mar 6. PMID 22390143
- [Result] Teo K, Lear S, Islam S, Mony P, Dehghan M, Li W, Rosengren A, Lopez-Jaramillo P, Diaz R, Oliveira G, Miskan M, Rangarajan S, Iqbal R, Ilow R, Puone T, Bahonar A, Gulec S, Darwish EA, Lanas F, Vijaykumar K, Rahman O, Chifamba J, Hou Y, Li N, Yusuf S; PURE Investigators. Prevalence of a healthy lifestyle among individuals with cardiovascular disease in high-, middle- and low-income countries: The Prospective Urban Rural Epidemiology (PURE) study. JAMA. 2013 Apr 17;309(15):1613-21. doi: 10.1001/jama.2013.3519. PMID 23592106
- [Result] Chow CK, Teo KK, Rangarajan S, Islam S, Gupta R, Avezum A, Bahonar A, Chifamba J, Dagenais G, Diaz R, Kazmi K, Lanas F, Wei L, Lopez-Jaramillo P, Fanghong L, Ismail NH, Puoane T, Rosengren A, Szuba A, Temizhan A, Wielgosz A, Yusuf R, Yusufali A, McKee M, Liu L, Mony P, Yusuf S; PURE (Prospective Urban Rural Epidemiology) Study investigators. Prevalence, awareness, treatment, and control of hypertension in rural and urban communities in high-, middle-, and low-income countries. JAMA. 2013 Sep 4;310(9):959-68. doi: 10.1001/jama.2013.184182. PMID 24002282
- [Result] Corsi DJ, Subramanian SV, Chow CK, McKee M, Chifamba J, Dagenais G, Diaz R, Iqbal R, Kelishadi R, Kruger A, Lanas F, Lopez-Jaramilo P, Mony P, Mohan V, Avezum A, Oguz A, Rahman MO, Rosengren A, Szuba A, Li W, Yusoff K, Yusufali A, Rangarajan S, Teo K, Yusuf S. Prospective Urban Rural Epidemiology (PURE) study: Baseline characteristics of the household sample and comparative analyses with national data in 17 countries. Am Heart J. 2013 Oct;166(4):636-646.e4. doi: 10.1016/j.ahj.2013.04.019. Epub 2013 Jul 27. PMID 24093842
- [Result] Duong M, Islam S, Rangarajan S, Teo K, O'Byrne PM, Schunemann HJ, Igumbor E, Chifamba J, Liu L, Li W, Ismail T, Shankar K, Shahid M, Vijayakumar K, Yusuf R, Zatonska K, Oguz A, Rosengren A, Heidari H, Almahmeed W, Diaz R, Oliveira G, Lopez-Jaramillo P, Seron P, Killian K, Yusuf S; PURE-BREATH Study Investigators. Global differences in lung function by region (PURE): an international, community-based prospective study. Lancet Respir Med. 2013 Oct;1(8):599-609. doi: 10.1016/S2213-2600(13)70164-4. Epub 2013 Sep 10. PMID 24461663
- [Result] Mahajan R, Malik M, Bharathi AV, Lakshmi PV, Patro BK, Rana SK, Kumar R. Reproducibility and validity of a quantitative food frequency questionnaire in an urban and rural area of northern India. Natl Med J India. 2013 Sep-Oct;26(5):266-72. PMID 25017832
- [Result] Mente A, O'Donnell MJ, Dagenais G, Wielgosz A, Lear SA, McQueen MJ, Jiang Y, Xingyu W, Jian B, Calik KB, Akalin AA, Mony P, Devanath A, Yusufali AH, Lopez-Jaramillo P, Avezum A Jr, Yusoff K, Rosengren A, Kruger L, Orlandini A, Rangarajan S, Teo K, Yusuf S. Validation and comparison of three formulae to estimate sodium and potassium excretion from a single morning fasting urine compared to 24-h measures in 11 countries. J Hypertens. 2014 May;32(5):1005-14; discussion 1015. doi: 10.1097/HJH.0000000000000122. PMID 24569420
- [Result] Lear SA, Teo K, Gasevic D, Zhang X, Poirier PP, Rangarajan S, Seron P, Kelishadi R, Tamil AM, Kruger A, Iqbal R, Swidan H, Gomez-Arbelaez D, Yusuf R, Chifamba J, Kutty VR, Karsidag K, Kumar R, Li W, Szuba A, Avezum A, Diaz R, Anand SS, Rosengren A, Yusuf S; Prospective Urban Rural Epidemiology (PURE) study. The association between ownership of common household devices and obesity and diabetes in high, middle and low income countries. CMAJ. 2014 Mar 4;186(4):258-66. doi: 10.1503/cmaj.131090. Epub 2014 Feb 10. PMID 24516093
- [Result] Mente A, O'Donnell MJ, Rangarajan S, McQueen MJ, Poirier P, Wielgosz A, Morrison H, Li W, Wang X, Di C, Mony P, Devanath A, Rosengren A, Oguz A, Zatonska K, Yusufali AH, Lopez-Jaramillo P, Avezum A, Ismail N, Lanas F, Puoane T, Diaz R, Kelishadi R, Iqbal R, Yusuf R, Chifamba J, Khatib R, Teo K, Yusuf S; PURE Investigators. Association of urinary sodium and potassium excretion with blood pressure. N Engl J Med. 2014 Aug 14;371(7):601-11. doi: 10.1056/NEJMoa1311989. PMID 25119606
- [Result] O'Donnell M, Mente A, Rangarajan S, McQueen MJ, Wang X, Liu L, Yan H, Lee SF, Mony P, Devanath A, Rosengren A, Lopez-Jaramillo P, Diaz R, Avezum A, Lanas F, Yusoff K, Iqbal R, Ilow R, Mohammadifard N, Gulec S, Yusufali AH, Kruger L, Yusuf R, Chifamba J, Kabali C, Dagenais G, Lear SA, Teo K, Yusuf S; PURE Investigators. Urinary sodium and potassium excretion, mortality, and cardiovascular events. N Engl J Med. 2014 Aug 14;371(7):612-23. doi: 10.1056/NEJMoa1311889. PMID 25119607
- [Result] Yusuf S, Rangarajan S, Teo K, Islam S, Li W, Liu L, Bo J, Lou Q, Lu F, Liu T, Yu L, Zhang S, Mony P, Swaminathan S, Mohan V, Gupta R, Kumar R, Vijayakumar K, Lear S, Anand S, Wielgosz A, Diaz R, Avezum A, Lopez-Jaramillo P, Lanas F, Yusoff K, Ismail N, Iqbal R, Rahman O, Rosengren A, Yusufali A, Kelishadi R, Kruger A, Puoane T, Szuba A, Chifamba J, Oguz A, McQueen M, McKee M, Dagenais G; PURE Investigators. Cardiovascular risk and events in 17 low-, middle-, and high-income countries. N Engl J Med. 2014 Aug 28;371(9):818-27. doi: 10.1056/NEJMoa1311890. PMID 25162888
- [Result] Batool S, O'Donnell M, Sharma M, Islam S, Dagenais GR, Poirier P, Lear SA, Wielgosz A, Teo K, Stotts G, McCreary CR, Frayne R, DeJesus J, Rangarajan S, Yusuf S, Smith EE; PURE Study Investigators. Incidental magnetic resonance diffusion-weighted imaging-positive lesions are rare in neurologically asymptomatic community-dwelling adults. Stroke. 2014 Jul;45(7):2115-7. doi: 10.1161/STROKEAHA.114.005782. Epub 2014 Jun 12. PMID 24923720
- [Result] Chow CK, Corsi DJ, Lock K, Madhavan M, Mackie P, Li W, Yi S, Wang Y, Swaminathan S, Lopez-Jaramillo P, Gomez-Arbelaez D, Avezum A, Lear SA, Dagenais G, Teo K, McKee M, Yusuf S. A novel method to evaluate the community built environment using photographs--Environmental Profile of a Community Health (EPOCH) photo neighbourhood evaluation tool. PLoS One. 2014 Nov 4;9(11):e110042. doi: 10.1371/journal.pone.0110042. eCollection 2014. PMID 25369366
- [Result] Smith EE, O'Donnell M, Dagenais G, Lear SA, Wielgosz A, Sharma M, Poirier P, Stotts G, Black SE, Strother S, Noseworthy MD, Benavente O, Modi J, Goyal M, Batool S, Sanchez K, Hill V, McCreary CR, Frayne R, Islam S, DeJesus J, Rangarajan S, Teo K, Yusuf S; PURE Investigators. Early cerebral small vessel disease and brain volume, cognition, and gait. Ann Neurol. 2015 Feb;77(2):251-61. doi: 10.1002/ana.24320. PMID 25428654
- [Result] Mayhew AJ, Lock K, Kelishadi R, Swaminathan S, Marcilio CS, Iqbal R, Dehghan M, Yusuf S, Chow CK. Nutrition labelling, marketing techniques, nutrition claims and health claims on chip and biscuit packages from sixteen countries. Public Health Nutr. 2016 Apr;19(6):998-1007. doi: 10.1017/S1368980015000658. Epub 2015 Mar 30. PMID 25818889
- [Result] Rosengren A, Teo K, Rangarajan S, Kabali C, Khumalo I, Kutty VR, Gupta R, Yusuf R, Iqbal R, Ismail N, Altuntas Y, Kelishadi R, Diaz R, Avezum A, Chifamba J, Zatonska K, Wei L, Liao X, Lopez-Jaramillo P, Yusufali A, Seron P, Lear SA, Yusuf S. Psychosocial factors and obesity in 17 high-, middle- and low-income countries: the Prospective Urban Rural Epidemiologic study. Int J Obes (Lond). 2015 Aug;39(8):1217-23. doi: 10.1038/ijo.2015.48. Epub 2015 Apr 14. PMID 25869608
- [Result] Leong DP, Teo KK, Rangarajan S, Lopez-Jaramillo P, Avezum A Jr, Orlandini A, Seron P, Ahmed SH, Rosengren A, Kelishadi R, Rahman O, Swaminathan S, Iqbal R, Gupta R, Lear SA, Oguz A, Yusoff K, Zatonska K, Chifamba J, Igumbor E, Mohan V, Anjana RM, Gu H, Li W, Yusuf S; Prospective Urban Rural Epidemiology (PURE) Study investigators. Prognostic value of grip strength: findings from the Prospective Urban Rural Epidemiology (PURE) study. Lancet. 2015 Jul 18;386(9990):266-73. doi: 10.1016/S0140-6736(14)62000-6. Epub 2015 May 13. PMID 25982160
- [Result] Gupta R, Islam S, Mony P, Kutty VR, Mohan V, Kumar R, Thakur JS, Shankar VK, Mohan D, Vijayakumar K, Rahman O, Yusuf R, Iqbal R, Shahid M, Mohan I, Rangarajan S, Teo KK, Yusuf S. Socioeconomic factors and use of secondary preventive therapies for cardiovascular diseases in South Asia: The PURE study. Eur J Prev Cardiol. 2015 Oct;22(10):1261-71. doi: 10.1177/2047487314540386. Epub 2014 Jun 18. PMID 24942224
- [Result] Smyth A, Teo KK, Rangarajan S, O'Donnell M, Zhang X, Rana P, Leong DP, Dagenais G, Seron P, Rosengren A, Schutte AE, Lopez-Jaramillo P, Oguz A, Chifamba J, Diaz R, Lear S, Avezum A, Kumar R, Mohan V, Szuba A, Wei L, Yang W, Jian B, McKee M, Yusuf S; PURE Investigators. Alcohol consumption and cardiovascular disease, cancer, injury, admission to hospital, and mortality: a prospective cohort study. Lancet. 2015 Nov 14;386(10007):1945-1954. doi: 10.1016/S0140-6736(15)00235-4. Epub 2015 Sep 17. PMID 26386538
- [Result] Savell E, Gilmore AB, Sims M, Mony PK, Koon T, Yusoff K, Lear SA, Seron P, Ismail N, Calik KB, Rosengren A, Bahonar A, Kumar R, Vijayakumar K, Kruger A, Swidan H, Gupta R, Igumbor E, Afridi A, Rahman O, Chifamba J, Zatonska K, Mohan V, Mohan D, Lopez-Jaramillo P, Avezum A, Poirier P, Orlandini A, Li W, McKee M, Rangarajan S, Yusuf S, Chow CK. The environmental profile of a community's health: a cross-sectional study on tobacco marketing in 16 countries. Bull World Health Organ. 2015 Dec 1;93(12):851-61G. doi: 10.2471/BLT.15.155846. PMID 26668437
- [Result] Lamelas PM, Mente A, Diaz R, Orlandini A, Avezum A, Oliveira G, Lanas F, Seron P, Lopez-Jaramillo P, Camacho-Lopez P, O Donnell MJ, Rangarajan S, Teo K, Yusuf S. Association of Urinary Sodium Excretion With Blood Pressure and Cardiovascular Clinical Events in 17,033 Latin Americans. Am J Hypertens. 2016 Jul;29(7):796-805. doi: 10.1093/ajh/hpv195. Epub 2015 Dec 18. PMID 26683344
- [Result] Khatib R, McKee M, Shannon H, Chow C, Rangarajan S, Teo K, Wei L, Mony P, Mohan V, Gupta R, Kumar R, Vijayakumar K, Lear SA, Diaz R, Avezum A, Lopez-Jaramillo P, Lanas F, Yusoff K, Ismail N, Kazmi K, Rahman O, Rosengren A, Monsef N, Kelishadi R, Kruger A, Puoane T, Szuba A, Chifamba J, Temizhan A, Dagenais G, Gafni A, Yusuf S; PURE study investigators. Availability and affordability of cardiovascular disease medicines and their effect on use in high-income, middle-income, and low-income countries: an analysis of the PURE study data. Lancet. 2016 Jan 2;387(10013):61-9. doi: 10.1016/S0140-6736(15)00469-9. Epub 2015 Oct 20. PMID 26498706
- [Result] Mente A, Dagenais G, Wielgosz A, Lear SA, McQueen MJ, Zeidler J, Fu L, DeJesus J, Rangarajan S, Bourlaud AS, De Bluts AL, Corber E, de Jong V, Boomgaardt J, Shane A, Jiang Y, de Groh M, O'Donnell MJ, Yusuf S, Teo K. Assessment of Dietary Sodium and Potassium in Canadians Using 24-Hour Urinary Collection. Can J Cardiol. 2016 Mar;32(3):319-26. doi: 10.1016/j.cjca.2015.06.020. Epub 2015 Jun 25. PMID 26454468
- [Result] Li W, Gu H, Teo KK, Bo J, Wang Y, Yang J, Wang X, Zhang H, Sun Y, Jia X, He X, Zhao X, Cheng X, Li J, Rangarajan S, Chen C, Yusuf S, Liu L; PURE China Investigators. Hypertension prevalence, awareness, treatment, and control in 115 rural and urban communities involving 47 000 people from China. J Hypertens. 2016 Jan;34(1):39-46. doi: 10.1097/HJH.0000000000000745. PMID 26630211
- [Result] Raina P, Sohel N, Oremus M, Shannon H, Mony P, Kumar R, Li W, Wang Y, Wang X, Yusoff K, Yusuf R, Iqbal R, Szuba A, Oguz A, Rosengren A, Kruger A, Chifamba J, Mohammadifard N, Darwish EA, Dagenais G, Diaz R, Avezum A, Lopez-Jaramillo P, Seron P, Rangarajan S, Teo K, Yusuf S; PURE Investigators. Assessing global risk factors for non-fatal injuries from road traffic accidents and falls in adults aged 35-70 years in 17 countries: a cross-sectional analysis of the Prospective Urban Rural Epidemiological (PURE) study. Inj Prev. 2016 Apr;22(2):92-8. doi: 10.1136/injuryprev-2014-041476. Epub 2015 Oct 28. PMID 26512093
- [Result] Leong DP, Teo KK, Rangarajan S, Kutty VR, Lanas F, Hui C, Quanyong X, Zhenzhen Q, Jinhua T, Noorhassim I, AlHabib KF, Moss SJ, Rosengren A, Akalin AA, Rahman O, Chifamba J, Orlandini A, Kumar R, Yeates K, Gupta R, Yusufali A, Dans A, Avezum A, Lopez-Jaramillo P, Poirier P, Heidari H, Zatonska K, Iqbal R, Khatib R, Yusuf S. Reference ranges of handgrip strength from 125,462 healthy adults in 21 countries: a prospective urban rural epidemiologic (PURE) study. J Cachexia Sarcopenia Muscle. 2016 Dec;7(5):535-546. doi: 10.1002/jcsm.12112. Epub 2016 Apr 12. PMID 27104109
- [Result] Dagenais GR, Gerstein HC, Zhang X, McQueen M, Lear S, Lopez-Jaramillo P, Mohan V, Mony P, Gupta R, Kutty VR, Kumar R, Rahman O, Yusoff K, Zatonska K, Oguz A, Rosengren A, Kelishadi R, Yusufali A, Diaz R, Avezum A, Lanas F, Kruger A, Peer N, Chifamba J, Iqbal R, Ismail N, Xiulin B, Jiankang L, Wenqing D, Gejie Y, Rangarajan S, Teo K, Yusuf S. Variations in Diabetes Prevalence in Low-, Middle-, and High-Income Countries: Results From the Prospective Urban and Rural Epidemiological Study. Diabetes Care. 2016 May;39(5):780-7. doi: 10.2337/dc15-2338. Epub 2016 Mar 10. PMID 26965719
- [Result] Mente A, O'Donnell M, Rangarajan S, Dagenais G, Lear S, McQueen M, Diaz R, Avezum A, Lopez-Jaramillo P, Lanas F, Li W, Lu Y, Yi S, Rensheng L, Iqbal R, Mony P, Yusuf R, Yusoff K, Szuba A, Oguz A, Rosengren A, Bahonar A, Yusufali A, Schutte AE, Chifamba J, Mann JF, Anand SS, Teo K, Yusuf S; PURE, EPIDREAM and ONTARGET/TRANSCEND Investigators. Associations of urinary sodium excretion with cardiovascular events in individuals with and without hypertension: a pooled analysis of data from four studies. Lancet. 2016 Jul 30;388(10043):465-75. doi: 10.1016/S0140-6736(16)30467-6. Epub 2016 May 20. PMID 27216139
- [Result] Miller V, Yusuf S, Chow CK, Dehghan M, Corsi DJ, Lock K, Popkin B, Rangarajan S, Khatib R, Lear SA, Mony P, Kaur M, Mohan V, Vijayakumar K, Gupta R, Kruger A, Tsolekile L, Mohammadifard N, Rahman O, Rosengren A, Avezum A, Orlandini A, Ismail N, Lopez-Jaramillo P, Yusufali A, Karsidag K, Iqbal R, Chifamba J, Oakley SM, Ariffin F, Zatonska K, Poirier P, Wei L, Jian B, Hui C, Xu L, Xiulin B, Teo K, Mente A. Availability, affordability, and consumption of fruits and vegetables in 18 countries across income levels: findings from the Prospective Urban Rural Epidemiology (PURE) study. Lancet Glob Health. 2016 Oct;4(10):e695-703. doi: 10.1016/S2214-109X(16)30186-3. Epub 2016 Aug 23. PMID 27567348
- [Result] Camacho PA, Gomez-Arbelaez D, Molina DI, Sanchez G, Arcos E, Narvaez C, Garcia H, Perez M, Hernandez EA, Duran M, Cure C, Sotomayor A, Rico A, David TM, Cohen DD, Rangarajan S, Yusuf S, Lopez-Jaramillo P. Social disparities explain differences in hypertension prevalence, detection and control in Colombia. J Hypertens. 2016 Dec;34(12):2344-2352. doi: 10.1097/HJH.0000000000001115. PMID 27662189
- [Result] Avezum A, Oliveira GBF, Lanas F, Lopez-Jaramillo P, Diaz R, Miranda JJ, Seron P, Camacho-Lopez PA, Orlandini A, Bernabe-Ortiz A, Cordeiro Mattos A, Islam S, Rangarajan S, Teo K, Yusuf S. Secondary CV Prevention in South America in a Community Setting: The PURE Study. Glob Heart. 2017 Dec;12(4):305-313. doi: 10.1016/j.gheart.2016.06.001. Epub 2016 Oct 20. PMID 27773540
- [Result] Palafox B, McKee M, Balabanova D, AlHabib KF, Avezum AJ, Bahonar A, Ismail N, Chifamba J, Chow CK, Corsi DJ, Dagenais GR, Diaz R, Gupta R, Iqbal R, Kaur M, Khatib R, Kruger A, Kruger IM, Lanas F, Lopez-Jaramillo P, Minfan F, Mohan V, Mony PK, Oguz A, Palileo-Villanueva LM, Perel P, Poirier P, Rangarajan S, Rensheng L, Rosengren A, Soman B, Stuckler D, Subramanian SV, Teo K, Tsolekile LP, Wielgosz A, Yaguang P, Yeates K, Yongzhen M, Yusoff K, Yusuf R, Yusufali A, Zatonska K, Yusuf S. Wealth and cardiovascular health: a cross-sectional study of wealth-related inequalities in the awareness, treatment and control of hypertension in high-, middle- and low-income countries. Int J Equity Health. 2016 Dec 8;15(1):199. doi: 10.1186/s12939-016-0478-6. PMID 27931255
- [Result] Duong M, Rangarajan S, Zhang X, Killian K, Mony P, Swaminathan S, Bharathi AV, Nair S, Vijayakumar K, Mohan I, Gupta R, Mohan D, Rani S, Mohan V, Iqbal R, Kazmi K, Rahman O, Yusuf R, Pinnaka LV, Kumar R, O'Byrne P, Yusuf S. Effects of bidi smoking on all-cause mortality and cardiorespiratory outcomes in men from south Asia: an observational community-based substudy of the Prospective Urban Rural Epidemiology Study (PURE). Lancet Glob Health. 2017 Feb;5(2):e168-e176. doi: 10.1016/S2214-109X(17)30004-9. PMID 28104186
- [Result] Gupta R, Kaur M, Islam S, Mohan V, Mony P, Kumar R, Kutty VR, Iqbal R, Rahman O, Deepa M, Antony J, Vijaykumar K, Kazmi K, Yusuf R, Mohan I, Panwar RB, Rangarajan S, Yusuf S. Association of Household Wealth Index, Educational Status, and Social Capital with Hypertension Awareness, Treatment, and Control in South Asia. Am J Hypertens. 2017 Apr 1;30(4):373-381. doi: 10.1093/ajh/hpw169. PMID 28096145
- [Result] Leong DP, McKee M, Yusuf S; PURE Investigators. Population Muscle Strength Predicts Olympic Medal Tallies: Evidence from 20 Countries in the PURE Prospective Cohort Study. PLoS One. 2017 Jan 20;12(1):e0169821. doi: 10.1371/journal.pone.0169821. eCollection 2017. PMID 28107362
- [Result] Khatib R, Giacaman R, Khammash U, Yusuf S. Challenges to conducting epidemiology research in chronic conflict areas: examples from PURE- Palestine. Confl Health. 2017 Feb 22;10:33. doi: 10.1186/s13031-016-0101-x. eCollection 2016. PMID 28239410
- [Result] Chow CK, Corsi DJ, Gilmore AB, Kruger A, Igumbor E, Chifamba J, Yang W, Wei L, Iqbal R, Mony P, Gupta R, Vijayakumar K, Mohan V, Kumar R, Rahman O, Yusoff K, Ismail N, Zatonska K, Altuntas Y, Rosengren A, Bahonar A, Yusufali A, Dagenais G, Lear S, Diaz R, Avezum A, Lopez-Jaramillo P, Lanas F, Rangarajan S, Teo K, McKee M, Yusuf S. Tobacco control environment: cross-sectional survey of policy implementation, social unacceptability, knowledge of tobacco health harms and relationship to quit ratio in 17 low-income, middle-income and high-income countries. BMJ Open. 2017 Mar 31;7(3):e013817. doi: 10.1136/bmjopen-2016-013817. PMID 28363924
- [Result] Yusufali AM, Khatib R, Islam S, Alhabib KF, Bahonar A, Swidan HM, Khammash U, Alshamiri MQ, Rangarajan S, Yusuf S. Prevalence, awareness, treatment and control of hypertension in four Middle East countries. J Hypertens. 2017 Jul;35(7):1457-1464. doi: 10.1097/HJH.0000000000001326. PMID 28486270
- [Derived] Chen R, Liu Y, Yang S, Lin Z, Yu G, Wang W, Wei D, Li W, Wang H, Zhang M, Zhang P, Zhang Y, Zhou F, Ding R. The prevalence, recognition, and treatment of depression and anxiety symptoms among Chinese cardiovascular outpatients. Sci Rep. 2025 Oct 21;15(1):36798. doi: 10.1038/s41598-025-20683-6. PMID 41120526
- [Derived] Narula N, Wong ECL, Mente A, Rangarajan S, Lang X, Li Q, Chen M, Mohan I, Mat-Nasir N, Diaz ML, Lopez-Jaramillo P, Bahonar A, Avezum A, Karsidag K, Rosengren A, Abat MEM, Lanas F, Swart EC, Yusuf R, Alhabib KF, Iqbal R, Basiak-Rasala A, Khatib R, Yusufali A, Yeates K, Chifamba J, Marshall JK, Moayyedi P, Reinisch W, Yusuf S. Ultraprocessed Grains and Risk of Inflammatory Bowel Disease: Results From the Prospective Urban Rural Epidemiology Study. Am J Gastroenterol. 2025 Aug 4. doi: 10.14309/ajg.0000000000003700. Online ahead of print. PMID 40758217
- [Derived] Joundi RA, Hu B, Rangarajan S, Leong DP, Islam S, Smith EE, Mirrakhimov E, Seron P, Alhabib KF, Assembekov B, Chifamba J, Yusuf R, Khatib R, Felix C, Yusufali A, Mohammadifard N, Rosengren A, Oguz A, Iqbal R, Yeates K, Avezum A, Kruger I, Anjana R, Pvm L, Gupta R, Zatonska K, Barbarash O, Pelliza E, Rammohan K, Li M, Li X, Ismail R, Lopez-Jaramillo P, Evans M, O'Donnell M, Yusuf S. Activity limitations, use of assistive devices, and mortality and clinical events in 25 high-income, middle-income, and low-income countries: an analysis of the PURE study. Lancet. 2024 Aug 10;404(10452):554-569. doi: 10.1016/S0140-6736(24)01050-X. Epub 2024 Jul 25. PMID 39068950
- [Derived] Walli-Attaei M, Rosengren A, Rangarajan S, Breet Y, Abdul-Razak S, Sharief WA, Alhabib KF, Avezum A, Chifamba J, Diaz R, Gupta R, Hu B, Iqbal R, Ismail R, Kelishadi R, Khatib R, Lang X, Li S, Lopez-Jaramillo P, Mohan V, Oguz A, Palileo-Villanueva LM, Poltyn-Zaradna K, R SP, Pinnaka LVM, Seron P, Teo K, Verghese ST, Wielgosz A, Yeates K, Yusuf R, Anand SS, Yusuf S; PURE investigators. Metabolic, behavioural, and psychosocial risk factors and cardiovascular disease in women compared with men in 21 high-income, middle-income, and low-income countries: an analysis of the PURE study. Lancet. 2022 Sep 10;400(10355):811-821. doi: 10.1016/S0140-6736(22)01441-6. PMID 36088949
- [Derived] Narula N, Wong ECL, Dehghan M, Mente A, Rangarajan S, Lanas F, Lopez-Jaramillo P, Rohatgi P, Lakshmi PVM, Varma RP, Orlandini A, Avezum A, Wielgosz A, Poirier P, Almadi MA, Altuntas Y, Ng KK, Chifamba J, Yeates K, Puoane T, Khatib R, Yusuf R, Bostrom KB, Zatonska K, Iqbal R, Weida L, Yibing Z, Sidong L, Dans A, Yusufali A, Mohammadifard N, Marshall JK, Moayyedi P, Reinisch W, Yusuf S. Association of ultra-processed food intake with risk of inflammatory bowel disease: prospective cohort study. BMJ. 2021 Jul 14;374:n1554. doi: 10.1136/bmj.n1554. PMID 34261638
- [Derived] Pertiwi K, Kupers LK, Geleijnse JM, Zock PL, Wanders AJ, Kruger HS, van Zyl T, Kruger IM, Smuts CM. Associations of linoleic acid with markers of glucose metabolism and liver function in South African adults. Lipids Health Dis. 2020 Jun 16;19(1):138. doi: 10.1186/s12944-020-01318-3. PMID 32546275
- [Derived] Dehghan M, Mente A, Rangarajan S, Mohan V, Lear S, Swaminathan S, Wielgosz A, Seron P, Avezum A, Lopez-Jaramillo P, Turbide G, Chifamba J, AlHabib KF, Mohammadifard N, Szuba A, Khatib R, Altuntas Y, Liu X, Iqbal R, Rosengren A, Yusuf R, Smuts M, Yusufali A, Li N, Diaz R, Yusoff K, Kaur M, Soman B, Ismail N, Gupta R, Dans A, Sheridan P, Teo K, Anand SS, Yusuf S. Association of egg intake with blood lipids, cardiovascular disease, and mortality in 177,000 people in 50 countries. Am J Clin Nutr. 2020 Apr 1;111(4):795-803. doi: 10.1093/ajcn/nqz348. PMID 31965140
- [Derived] Wentzel-Viljoen E, Laubscher R, Vorster HH. Changes in food intake from 2005 to 2010 by a cohort of black rural and urban African men and women in the North West Province of South Africa: the PURE-NWP-SA study. Public Health Nutr. 2018 Nov;21(16):2941-2958. doi: 10.1017/S1368980018001878. Epub 2018 Aug 28. PMID 30149823
- [Derived] Wentzel-Viljoen E, Lee S, Laubscher R, Vorster HH. Accelerated nutrition transition in the North West Province of South Africa: results from the Prospective Urban and Rural Epidemiology (PURE-NWP-SA) cohort study, 2005 to 2010. Public Health Nutr. 2018 Oct;21(14):2630-2641. doi: 10.1017/S1368980018001118. Epub 2018 May 8. PMID 29734966
- See also: Study Webpage — http://www.phri.ca/pure/